CLINICAL TRIAL: NCT04407286
Title: Vitamin D Testing and Treatment for Adults With COVID 19
Brief Title: Vitamin D Testing and Treatment for COVID 19
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Arizona State University (Other)
Collaborators: Southwest College of Naturopathic Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00011960
Record Dates: First submitted 2020-05-19; First posted 2020-05-29 (Actual); Last update posted 2021-12-30 (Actual); Status verified 2021-12

CONDITIONS: Covid 19; Vitamin D Deficiency
MeSH Terms: conditions — COVID-19; Vitamin D Deficiency | interventions — Cholecalciferol

STUDY DESIGN:
Intervention Model Description: This is an open label treatment study for people with COVID 19 and low levels of vitamin D
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Group (Experimental): This group will receive vitamin D.
  The dosage for the first two weeks will be 10,000 IU/day b.i.d. (age 18-69 years) or 15,000 IU/day t.i.d. (age 70+)
  After two weeks of taking vitamin D, if vitamin D levels are still below 30 ng/ml, continue the dosage for 3 more weeks. If vitamin D levels are 30-49 ng/ml, continue at a dosage of 5000 IU/day. If vitamin D levels are 50+ ng/ml, stop supplementation.
  Interventions: Dietary Supplement: Vitamin D3

INTERVENTIONS:
Dietary Supplement: Vitamin D3 — Oral vitamin D3 capsules

SUMMARY:
This study will measure vitamin D levels in adults with COVID 19. Participants with low levels of vitamin D will be entered into an open label trial of supplementation with vitamin D.

DETAILED DESCRIPTION:
Protocol for Part 1:

* A single blood draw at SCNM to measure levels of vitamin D and other nutrients, comprehensive metabolic panel, and complete blood count with differential
* Completing a medical history/symptom form
* Completing a form about COVID-19 symptoms every 2 weeks for 6 weeks
* Authorization for release of medical records related to COVID 19 testing and/or treatment.

Protocol for Part 2:

* Take a vitamin D supplement daily for two weeks, at a dosage of 10,000 IU/day b.i.d. (age 18-69 years) or 15,000 IU/day t.i.d. (age 70+)
* After two weeks of taking vitamin D, return to SCNM for a blood draw to remeasure levels of vitamin D, comprehensive metabolic panel, and complete blood count with differential. If vitamin D levels are still below 30 ng/ml, continue the dosage for 3 more weeks. If vitamin D levels are 30-49 ng/ml, continue at a dosage of 5000 IU/day. If vitamin D levels are 50+ ng/ml, stop supplementation.
* Completing questionnaires about COVID 19 symptoms at 2, 4, and 6 weeks after treatment begins (5 minutes each time).

ELIGIBILITY:
Inclusion Criteria for Part 1 (testing):

1. Adult age 18 or older
2. Previous positive test result for COVID 19
3. Able to communicate clearly in English Exclusion Criteria for Part 1 (testing): none

Inclusion Criteria for Part 2 (Vitamin D supplementation)

1. Participation in Part 1
2. Vitamin D level below 30 ng/ml
3. No abnormalities on the comprehensive metabolic panel that are clinically significant to increasing the risk of an adverse reaction to vitamin D supplementation

Exclusion Criteria for Part 2 (Vitamin D supplementation):

1. Liver impairment
2. Clinical opinion of study physician that vitamin D supplementation could be harmful to the participant.
3. Pregnancy
4. No symptoms for 2 weeks after positive COVID 19 test
5. Recovered from symptoms

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2020-05-19 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Vitamin D levels | baseline and after two weeks of vitamin D supplementation
  change in level of Vitamin D, 25-Hydroxy between the two time points
severity of COVID 19 symptoms | baseline and at 2 weeks after vitamin D supplementation
  We will calculate the change in severity of COVID 19 symptoms from baseline to 2 weeks after vitamin D supplementation

CONTACTS AND LOCATIONS:
Overall Officials: James B Adams, PhD, Principal Investigator — Arizona State University; Sarah Trahan, NMD, Principal Investigator — Southwest College of Naturopathic Medicine
Locations (1):
- Arizona State University, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: Undecided
Contact us if you wish to discuss sharing of de-identified data